CLINICAL TRIAL: NCT01423578
Title: Effects of Yoga and Cardiovascular Exercise on Smoking Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-15245
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Tobacco Dependence
Keywords: craving; mood; cue reactivity; smoking behavior; quit smoking; prevention; Hatha yoga; cardiovascular exercise
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Yoga; Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hatha Yoga (HY) (Active Comparator): Exercise and Smoking Cessation Counseling
  Interventions: Behavioral: Hatha Yoga (HY); Behavioral: Smoking Cessation Counseling
- Cardiovascular Exercise (CE) (Experimental): Exercise and Smoking Cessation Counseling
  Interventions: Behavioral: Cardiovascular Exercise (CE); Behavioral: Smoking Cessation Counseling
- Smoking Cessation Counseling Only (Other): Control Group - Smoking Cessation Counseling
  Interventions: Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Behavioral: Hatha Yoga (HY) — 3 Sessions of yoga instruction
  Other Names: yoga
  Arms: Hatha Yoga (HY)
Behavioral: Cardiovascular Exercise (CE) — 3 sessions of cardiovascular exercise
  Other Names: exercise
  Arms: Cardiovascular Exercise (CE)
Behavioral: Smoking Cessation Counseling — 4 smoking cessation counseling visits.
  Other Names: control group

SUMMARY:
The overall purpose of this pilot study is to examine effects of Hatha yoga and cardiovascular exercise on craving, mood, cue reactivity, and smoking behavior. Our preliminary study indicated that a single session of either form of activity intervention improved mood, and the yoga intervention appeared to decrease cravings to smoke. The proposed study will extend this preliminary research in several ways.

DETAILED DESCRIPTION:
First, the investigators will expand the exercise-based interventions from one to three sessions, which will more closely resemble how these interventions may be used in the context of smoking cessation. Second, the investigators will recruit smokers who are motivated to quit smoking, further increasing the clinical relevance of the research. Finally, the investigators will examine the effects of the interventions on actual smoking behavior within and outside of the laboratory setting. This may appropriately be considered a "proof of concept" study, as the investigators will not be powered to detect treatment outcome (smoking cessation) differences, nor are the interventions designed to maximize clinical smoking cessation outcomes.

Participants will be randomized to receive 3-sessions of yoga instruction, 3-sessions of cardiovascular exercise, or to a no activity control group. Sessions will be scheduled to occur approximately 7 days apart, with a minimum of 4 between sessions. Mood and craving will be assessed before and after each session, and smoking behavior will be assessed following each session. Finally, a detailed cue reactivity assessment will be conducted prior to the first session and following the last session. Analyses will examine intervention effects on craving, mood, cue reactivity, and smoking behavior. In addition, the investigators will examine several potential mediators and moderators of intervention effects on smoking behavior. Finally, the investigators will continue to examine the feasibility and potential acceptability of each active intervention, to assist in developing future clinical applications of these techniques in the context of smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 10 cigarettes per day
* Smoked regularly at least 2 years
* Carbon monoxide reading at least 8 ppm
* Interest in quitting smoking
* Able to read and understand the consent form and questionnaires
* Not currently practicing yoga

Exclusion Criteria:

* Current Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) (American Psychiatric Association, 1994) psychosis
* Major depressive episode, manic episode, or panic disorder
* Current DSM-IV psychoactive substance dependence or use
* Current medication use that might affect physiological responses
* Current use of bupropion, varenicline, or nicotine-containing products other than cigarettes
* Significant health problems that might compromise physiological data collection or be contraindicated for moderate physical exercise or yoga
* Significant hearing or visual impairment; pregnant as determined by urine human chorionic gonadotropin (hCG) test or nursing females
* Body mass index (BMI) 35 or greater

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2007-08-21 (Actual); Primary Completion 2011-05-02 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
The Number of Participants Reporting Post Intervention Effects | Average of 6 Months
  Intervention effects on measures of craving, mood, cue reactivity, and smoking behavior will be analyzed with mixed-design analysis of variance (ANOVA), with Intervention as the between-group factor (HY vs. CE vs. NA), and Time as a within-subject factor (pre vs. post-intervention). Analyses for cue reactivity variables will include the additional within-subject factor of Cue Type (smoking vs. neutral), and analyses for craving and mood self-report will include the additional within-subject factor of Session (1 vs. 2 vs. 3).

SECONDARY OUTCOMES:
Number of Participants Reporting Behavior Changes Post Intervention | Average of 6 Months
  In order to determine whether intervention effects on smoking behavior are mediated by changes in craving, mood, and/or cue reactivity, we will conduct Sobel tests (e.g., Preacher & Leonardelli, 2001), supplemented by mediation analyses using methods of Baron & Kenny (1986).

CONTACTS AND LOCATIONS:
Overall Officials: David J. Drobes, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States